CLINICAL TRIAL: NCT04865770
Title: Renal Mode of Action of Semaglutide in Patients With Type 2 Diabetes and Chronic Kidney Disease
Brief Title: A Research Study to Find Out How Semaglutide Works in the Kidneys Compared to Placebo, in People With Type 2 Diabetes and Chronic Kidney Disease (the REMODEL Trial)
Acronym: REMODEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4662; U1111-1248-7912 (Other: World Health Organization (WHO)); 2020-000828-19 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide 1.0 mg OW (Experimental): Once-weekly (OW) Semaglutide administered subcutaneously (s.c., under the skin).
  Interventions: Drug: Semaglutide
- Placebo (Semaglutide) 1.0 mg OW (Placebo Comparator): Once-weekly (OW) placebo (Semaglutide) administered subcutaneously (s.c., under the skin).
  Interventions: Drug: Placebo (Semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide given subcutaneously (sc, under the skin) once weekly. Dose gradually increased over 8 weeks from 0.25 to 1.0 mg. The study will last for about 1 year.
  Arms: Semaglutide 1.0 mg OW
Drug: Placebo (Semaglutide) — Placebo (Semaglutide) given subcutaneously (sc, under the skin) once weekly. Dose gradually increased over 8 weeks from 0.25 to 1.0 mg. The study will last for about 1 year.
  Arms: Placebo (Semaglutide) 1.0 mg OW

SUMMARY:
We are doing this study to learn more about how semaglutide may help fight chronic kidney disease in people with type 2 diabetes. We are doing this by looking into how semaglutide works in the kidneys.

Participants will either get semaglutide or placebo (a 'dummy' medicine) - which treatment participants get is decided by chance.

Semaglutide is a medicine doctors can prescribe in some countries for the treatment of type 2 diabetes.

Participants will get the study medicine in a pen. Participants will use the pen to inject the medicine into the skin once a week.

The study will last for about 1 year. Participants will have 11 visits to the clinic, and 2 phone visits. Some of the visits could be in different locations.

Study staff will take blood samples at most of these visits. At 9 visits, participants will be asked to bring a sample of their first morning urine. At 4 of the visits participants will have to bring urine that they have collected over the last 24 hours.

The study includes magnetic resonance imaging (MRI) scans of participants' kidneys which is a test that shows a detailed picture of organs and other parts inside the body. The scan will last for 30 minutes, and is free of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with T2D (type 2 diabetes) greater than or equal to 180 days prior to the day of screening.
* HbA1c (glycated haemoglobin) below or equal to 9.0 percent (below or equal to 75 mmol/mol).
* Depending on biopsy/non-biopsy population:

  1. For subjects in the non-biopsy population: Serum creatinine-based eGFR greater than or equal to 30 and below or equal to 75 mL/min/1.73 m^2(CKD-EPI).
  2. For subjects in the biopsy sub-population: Serum creatinine-based eGFR greater than or equal to 40 and below or equal to 75 mL/min/1.73 m^2(CKD-EPI).
* UACR ( Urinary albumin-to-creatinine ratio ) greater than or equal to 20 and below 5000 mg/g.
* Treatment with maximum labelled or tolerated dose of a renin-angiotensin-aldosterone system (RAAS) blocking agent including an angiotensin converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB)) unless such treatment is contraindicated or not tolerated.Treatment dose must be stable for at least 28 days prior to screening.

Exclusion Criteria:

* Use of any glucagon-like peptide 1 receptor agonist (GLP-1 RA) within 30 days prior to screening.
* A prior solid organ transplant or awaiting solid organ transplant.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Presence or history of malignant neoplasms (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) within 5 years prior to the day of screening.
* Congenital or hereditary kidney diseases including polycystic kidney disease, autoimmune kidney diseases including glomerulonephritis or congenital urinary tract malformations.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and Visit 2. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Treatment with systemic anti-inflammatory or immunosuppressant drugs within 90 days prior to screening. Stable treatment with acetylsalicylic acid for prevention of cardiovascular events and occasional use of propionic acid derivatives drugs (e.g. ibuprofen) is allowed.
* Any contraindication for MRI according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
* Combination use of an ACE (angiotensin-converting enzyme) inhibitor and an ARB (angiotensin II receptor blockers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept.2834), Study Director — Novo Nordisk A/S
Locations (49):
- United States (20):
  - University of Arizona-CaTs, Tucson, Arizona
  - Academic Medical Research Institute, Los Angeles, California
  - Roderick A. Comunale II MD Inc., National City, California
  - N America Res Inst - San Dimas, San Dimas, California
  - UC Anschutz Medical Campus, Aurora, Colorado
  - Advent Health-Res Inst, Orlando, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University Hsptl - Atlanta, Atlanta, Georgia
  - Endeavor Health Glenbook Hosp, Evanston, Illinois
  - North Suburban Nephrology LLC, Gurnee, Illinois
  - University of Minnesota Health Clinical, Minneapolis, Minnesota
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Cleveland Clinic_Cleveland, Cleveland, Ohio
  - Prolato Clinical Research Cntr, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - University of Texas San Antonio, San Antonio, Texas
  - Univ of Washington Med Ctr, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
- Denmark (3):
  - Nefrologisk Klinik P 2132, Copenhagen
  - Rigshospitalet - Nefrologisk Klinik P 2132, Copenhagen
  - Steno Diabetes Center Copenhagen, Herlev
- France (6):
  - Centre Hospitalier Universitaire Amiens Picardie-Site Sud, Amiens
  - Centre Hospitalier Universitaire de Rouen - Hopital de Bois Guillaume, Bois-Guillaume
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-2, Grenoble - Cédex 09
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Chu de Reims-Hopital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil, Toulouse
- Italy (5):
  - Istituto Scientifico San Raffaele, Milan, MI
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera di Padova Clin.Med.3, Padua
  - Presidio Ospedaliero Cisanello, Pisa
  - Azienda Ospedaliero - Universitaria Sant'Andrea, Roma
- Poland (5):
  - In-Vivo Sp. z o.o., Bydgoszcz
  - Centrum Medyczne "Diabetika", Radom
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM W Szczecinie, Szczecin
  - Miedzyleski Szpital Specjalistyczny, Oddzial Nefrologiczny, Warsaw
  - Prywatny Gabinet Janusz Gumprecht, Zabrze
- South Africa (4):
  - Maxwell Centre, Durban, KwaZulu-Natal
  - Precise Clinical Solutions (Pty) Ltd, Durban, KwaZulu-Natal
  - Lenmed Shifa Private Hospital, Durban, KwaZulu-Natal
  - Prof Rayner_Division of Nephrology, Cape Town, Western Cape
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Pruijm M, Belmar N, Bjornstad P, Cherney DZI, Das V, Gunnarsson T, Hodgin JB, Schytz PA, Tuttle KR, Kretzler M. REMODELing mechanistic trials for kidney disease: a multimodal, tissue-centered approach to understand the renal mechanism of action of semaglutide. Kidney Int. 2026 Jan;109(1):6-16. doi: 10.1016/j.kint.2025.10.005. Epub 2025 Nov 7. PMID 41207620
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Mendonca L, Moura H, Chaves PC, Neves JS, Ferreira JP. The Impact of Glucagon-Like Peptide-1 Receptor Agonists on Kidney Outcomes: A Meta-Analysis of Randomized Placebo-Controlled Trials. Clin J Am Soc Nephrol. 2024 Oct 8;20(2):159-68. doi: 10.2215/CJN.0000000584. Online ahead of print. PMID 39480988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 31 sites in 8 countries.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive semaglutide or placebo, respectively. Both added to standard-of-care treatment.
Groups:
- Semaglutide 1.0 mg: Participants received once-weekly (OW) subcutaneous (s. c.) injection of semaglutide for 52 weeks. Participants received a dose of 0.25 milligrams (mg) from week 0 to week 4, then the dose was increased to 0.5 mg from week 4 to week 8. From week 8 to week 52, the dosage was 1.0 mg.
- Placebo: Participants received once-weekly (OW) subcutaneous injection (s. c.) of placebo matched for semaglutide for 52 weeks.
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Placebo
Started | 71 | 35
Full Analysis Set | 71 | 35
Safety Analysis Set | 71 | 35
Completed | 58 | 34
Not Completed | 13 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 9 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Placebo | Total
Number analyzed (Participants) | 71 | 35 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.2) | 65.1 (11.3) | 65.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 55 | 26 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 59 | 28 | 87
  Unknown or Not Reported | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 2 | 0 | 2
  Black Or African American | 5 | 5 | 10
  Not Reported | 6 | 4 | 10
  White | 43 | 22 | 65
  Other | 4 | 0 | 4
  Asian | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Kidney Oxygenation (Cortex), Blood Oxygenation-level Dependent Magnetic Resonance Imaging (BOLD MRI) (R2*)
Description: Change in kidney oxygenation in cortex assessed by BOLD (blood oxygenation level dependent) MRI from baseline (week 0) to end of treatment (week 52) is presented. R2* is a measure used in BOLD MRI to indicate the level of tissue oxygenation. A higher R2* value means lower tissue oxygenation while a lower R2* value means higher tissue oxygenation.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: Full analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product. Overall number of participants analyzed= FAS. Number Analyzed= number of participants with available data for particular timepoint, for the respective arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of kidney oxygenation (cortex)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of kidney oxygenation (cortex)
  Bilateral cortex: number analyzed (Participants) | 58 | 33
  Bilateral cortex | 0.98 (5.35) | 1.00 (7.39)
  Right cortex: number analyzed (Participants) | 58 | 33
  Right cortex | 0.98 (5.65) | 0.99 (7.26)
  Left cortex: number analyzed (Participants) | 58 | 31
  Left cortex | 0.98 (7.51) | 1.01 (9.12)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Bilateral cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate, on log scale; Test type: Other; p = 0.1333, ANCOVA; Treatment ratio = 0.98, 95% CI 2-sided [0.96 to 1.01]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; Right cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate, on log scale; Test type: Other; p = 0.2487, ANCOVA; Treatment ratio = 0.99, 95% CI 2-sided [0.96 to 1.01]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Placebo; Left cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate, on log scale; Test type: Other; p = 0.0907, ANCOVA; Treatment ratio = 0.97, 95% CI 2-sided [0.94 to 1.00]

2. Primary Outcome: Change in Kidney Oxygenation (Medulla), BOLD MRI (R2*)
Description: Change in kidney oxygenation in medulla assessed by BOLD (blood oxygenation level dependent) MRI from baseline (week 0) to end of treatment (week 52) is presented. R2* is a measure used in BOLD MRI to indicate the level of tissue oxygenation. A higher R2* value means lower tissue oxygenation while a lower R2* value means higher tissue oxygenation.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of kidney oxygenation (medulla)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of kidney oxygenation (medulla)
  Bilateral medulla: number analyzed (Participants) | 57 | 33
  Bilateral medulla | 0.99 (8.97) | 1.01 (11.37)
  Right medulla: number analyzed (Participants) | 57 | 33
  Right medulla | 0.98 (10.09) | 1.02 (10.83)
  Left medulla: number analyzed (Participants) | 58 | 31
  Left medulla | 0.99 (10.25) | 1.02 (13.02)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Bilateral medulla: The responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.5619, ANCOVA; Treatment ratio = 0.99, 95% CI 2-sided [0.94 to 1.03]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; Right medulla: The responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.2774, ANCOVA; Treatment ratio = 0.97, 95% CI 2-sided [0.93 to 1.02]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Placebo; Left medulla: The responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.7924, ANCOVA; Treatment ratio = 0.99, 95% CI 2-sided [0.94 to 1.04]

3. Primary Outcome: Change in Global Kidney Perfusion (MRI)
Description: Change in global kidney perfusion assessed by phase contrast MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of global kidney perfusion
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of global kidney perfusion
  Bilateral kidney: number analyzed (Participants) | 49 | 30
  Bilateral kidney | 1.03 (26.43) | 0.99 (24.39)
  Right kidney: number analyzed (Participants) | 50 | 30
  Right kidney | 1.04 (27.84) | 0.98 (28.85)
  Left kidney: number analyzed (Participants) | 50 | 29
  Left kidney | 1.02 (29.25) | 1.01 (26.83)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Bilateral kidney: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.0958, ANCOVA; Treatment ratio = 1.10, 95% CI 2-sided [0.98 to 1.24]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; Right kidney: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.0145, ANCOVA; Treatment ratio = 1.17, 95% CI 2-sided [1.03 to 1.33]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Placebo; Left kidney: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.3311, ANCOVA; Treatment ratio = 1.06, 95% CI 2-sided [0.94 to 1.21]

4. Primary Outcome: Change in Kidney Inflammation (Cortex), Longitudinal Relaxation Time (T1) Mapping (MRI)
Description: Change in kidney inflammation in cortex assessed by T1 mapping MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of kidney inflammation (cortex)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of kidney inflammation (cortex)
  Bilateral cortex: number analyzed (Participants) | 56 | 32
  Bilateral cortex | 1.01 (3.78) | 1.01 (5.43)
  Right cortex: number analyzed (Participants) | 56 | 32
  Right cortex | 1.01 (3.88) | 1.01 (5.57)
  Left cortex: number analyzed (Participants) | 56 | 31
  Left cortex | 1.01 (3.93) | 1.01 (5.71)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Bilateral cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.8651, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; Right cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.7240, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Placebo; Left cortex: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.7195, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.02]

5. Primary Outcome: Change in Kidney Inflammation (Medulla), T1 Mapping (MRI)
Description: Change in kidney inflammation in medulla assessed by T1 mapping MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of kidney inflammation (medulla)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of kidney inflammation (medulla)
  Bilateral medulla: number analyzed (Participants) | 56 | 32
  Bilateral medulla | 1.00 (3.56) | 1.00 (5.13)
  Right medulla: number analyzed (Participants) | 56 | 32
  Right medulla | 1.00 (3.90) | 1.01 (4.85)
  Left medulla: number analyzed (Participants) | 56 | 31
  Left medulla | 1.00 (3.69) | 1.00 (5.91)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Placebo; Bilateral medulla: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.9335, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; Right medulla: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.6517, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 3: Comparison: Semaglutide 1.0 mg vs Placebo; Left medulla: Responses are analysed using an ANCOVA with actual treatment, region and the stratification factors as categorical effects and the baseline value as a covariate; Test type: Other; p = 0.9017, ANCOVA; Treatment ratio = 1.00, 95% CI 2-sided [0.98 to 1.02]

6. Secondary Outcome: Change in Gene Expression Assessed by Single Nucleus Ribonucleic Acid (RNA) Sequencing (Kidney Biopsy)
Description: Changes in gene expression were assessed by single nucleus RNA sequencing (kidney biopsies) from baseline (week 0) to end of treatment (week 52). Cell type annotation was performed prior to the analysis. The analysis reports the log2 fold change in form of differential gene expression per cell type from baseline, comparing treatment arms. Genes are considered significant if fold change > 0.5 or < 0.5 and false discovery rate (FDR) <0.1; these criteria help identify biologically significant genes that are reliably differentially expressed in patients with conditions such as Type 2 diabetes and chronic kidney disease. The differential expression was estimated using a linear mixed model that included participant as a random effect. The cell types presented are those that contain these differentially expressed genes demonstrating the treatment response. This threshold is based on findings published in cross-sectional observational studies related to disease impact and gene activity.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: Full analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product. Overall Number participants analyzed = number of participants with available data for particular timepoint, for the respective arms.
Measure: Number; unit: log2 fold-change
Groups:
- Semaglutide 1.0 mg/Placebo: Participants received OW treatment with 0.25 mg semaglutide or placebo from week 0 to week 4 followed by 0.5 mg semaglutide or placebo from week 4 to week 8 followed by 1 mg semaglutide or placebo from week 8 to week 52 depending on the arm they were randomised to. This arm has combined data from Semaglutide arm and Placebo arm.
Arm/Group | Semaglutide 1.0 mg/Placebo
Number analyzed (Participants) | 22
log2 fold-change
  CNT-2, RSPO3 | 3.468216523
  CNT-Immune, SLC8A1-AS1 | 2.8531071
  EC-GC-1, KCNK6 | -1.952545192
  EC-GC-1, EMC10 | -2.485824696
  EC-GC-1, ENSG00000286145 | 1.831300888
  EC-GC-1, LMF1 | -1.528463786
  EC-GC-1, ANKUB1 | 1.783402404
  EC-GC-1, AHNAK | -1.368952211
  EC-GC-1, ENSG00000286150 | 1.318309657
  EC-GC-1, NSUN6 | -1.464540152
  EC-GC-1, TFCP2L1 | -2.24516792
  EC-GC-1, ENSG00000274422 | -1.860725608
  EC-GC-1, DPYD-AS1 | 1.996950045
  EC-GC-1, ENSG00000248138 | 2.110414741
  EC-GC-1, ACSM2B | -1.785467699
  EC-GC-1, CCNH | 1.033873239
  EC-GC-1, QTRT1 | -2.415240141
  EC-GC-1, CROCCP3 | -1.254541813
  EC-GC-1, ENSG00000251034 | 1.750285729
  EC-GC-1, LSAMP | -2.439268964
  EC-GC-1, LHX1-DT | -4.256689925
  EC-GC-1, ESRRG | -1.527414037
  EC-GC-1, CNTNAP2 | -2.377391827
  EC-GC-1, ENSG00000284966 | 1.665764749
  EC-GC-1, BICC1 | -1.445239386
  EC-GC-1, GNA14-AS1 | 1.192645521
  EC-GC-1, GUSBP11 | -1.318511642
  EC-GC-1, ENSG00000233783 | 1.668536087
  EC-GC-1, SEMA6A-AS1 | 1.183886707
  EC-GC-1, RBMS3-AS2 | 1.572052032
  EC-GC-1, ENSG00000286147 | -4.468841041
  EC-GC-1, LINC00342 | -1.151143461
  EC-GC-1, IRF3 | -1.566408786
  EC-GC-1, ENSG00000249207 | 1.35685803
  EC-GC-1, CRADD-AS1 | 1.972404772
  EC-GC-1, TOX3 | -2.206055055
  EC-GC-1, ENSG00000286458 | 1.271036656
  EC-GC-1, SLC12A3 | -2.531722898
  EC-GC-1, TALAM1 | 1.235573321
  EC-GC-1, PCDH17 | 1.107442597
  EC-GC-1, ATP13A3 | 1.078246118
  EC-GC-1, ENSG00000231772 | -2.382264501
  EC-GC-1, FBXL19 | -2.166973377
  EC-GC-1, ENSG00000254420 | 1.74612131
  EC-GC-1, SPC25 | 1.329461228
  EC-GC-1, SMAD4 | 1.13655744
  EC-GC-1, UFM1 | 1.20264148
  EC-GC-1, ENSG00000259564 | 2.071724947
  EC-GC-1, SHOC1 | 1.634369451
  EC-GC-1, MEF2C-AS2 | 1.753288691
  EC-GC-1, ENSG00000285801 | 1.440844025
  EC-GC-1, FAM228B | -1.22996414
  EC-GC-1, GLS | 0.868999317
  EC-GC-1, GDPD4 | -6.564026305
  EC-GC-1, INSYN2A | 1.759769032
  EC-GC-1, TNFRSF14 | -1.254004029
  EC-GC-1, PRX | -1.199880651
  EC-GC-1, PNN | -1.024604708
  EC-GC-1, KCNQ1OT1 | -0.794847103
  EC-GC-1, ACAP3 | -1.44397269
  EC-GC-1, BASP1-AS1 | -4.83539932
  EC-GC-1, RBFOX1 | -1.706411849
  EC-GC-1, CCDC90B-AS1 | -1.678217382
  EC-GC-1, ENSG00000240499 | 1.514399208
  EC-GC-1, LINC03076 | 1.545248095
  EC-GC-1, LINC01409 | -1.022992954
  EC-GC-1, CCT4 | 1.455396063
  EC-GC-1, CDC73 | 0.802691458
  EC-GC-1, NUMA1 | -0.931923316
  EC-GC-1, FLT4 | -0.935590968
  EC-GC-1, PDLIM5 | 0.764926487
  EC-GC-1, SPCS3 | 1.02068757
  EC-GC-1, ENSG00000250646 | 1.917331079
  EC-GC-1, ENSG00000258168 | 1.083991656
  EC-GC-1, ST8SIA4 | 0.901071433
  EC-GC-1, BCL2L1-AS1 | 1.262413164
  EC-GC-1, NRSN2-AS1 | -1.275348201
  EC-GC-1, STARD13-AS | 1.148054491
  EC-GC-1, CFLAR-AS1 | 1.168941896
  EC-GC-1, PRKAR1A | 1.257792414
  EC-GC-1, ENSG00000226239 | 1.126077043
  EC-GC-1, CTNNA3 | -1.819759686
  EC-GC-1, KCNK5 | -2.491597199
  EC-GC-1, ESR2 | 1.071576206
  EC-GC-1, SLC25A46 | 1.062235788
  EC-GC-1, REV3L | 0.792446528
  EC-GC-1, ZC2HC1C | 2.027909336
  EC-GC-1, ENSG00000279686 | -1.453758633
  EC-GC-1, ACER1 | -5.256214457
  EC-GC-1, MALRD1 | -2.36001857
  EC-GC-1, RRBP1 | -0.837125744
  EC-GC-1, ZNF451-AS1 | 1.853753635
  EC-GC-1, SHANK2 | -1.481833304
  EC-GC-1, ENSG00000248388 | 2.196067138
  EC-GC-1, KPNA5 | 0.936135624
  EC-GC-1, APPAT | -1.750949862
  EC-GC-1, PCNT | -0.932423432
  EC-GC-1, ENSG00000233848 | 2.752498803
  EC-GC-1, MORF4L2 | 1.28059543
  EC-GC-1, ENSG00000236283 | -1.572597604
  EC-GC-1, SNRNP70 | -0.883484114
  EC-GC-1, EXD3 | -0.805539835
  EC-GC-1, CNTNAP5 | -2.392758482
  EC-GC-1, CASR | -2.323412555
  EC-GC-1, ENSG00000285692 | 1.124516569
  EC-GC-1, WDR81 | -2.102548546
  EC-GC-1, ZNF160 | -0.907890266
  EC-GC-1, CA12 | -1.63720477
  EC-GC-1, MAPK8IP3 | -0.998528168
  EC-GC-1, ABTB3 | -2.945080572
  EC-GC-1, CHORDC1 | 1.047593755
  EC-GC-1, FREM1 | -1.948982139
  EC-GC-1, FXYD6-AS1 | 2.22442108
  EC-GC-1, SPACA6 | -1.045439073
  EC-GC-1, AGBL1 | -2.851170905
  EC-GC-2, NES | -2.451444521
  EC-GC-2, ADARB2 | -3.212266234
  EC-GC-2, SERPINB9 | 2.315559798
  EC-GC-2, ENSG00000274422 | -2.329265154
  EC-GC-2, BTNL9 | -2.01168798
  EC-GC-2, CPEB2 | 1.51543417
  EC-GC-2, TBX2 | -2.604511077
  EC-GC-2, ENSG00000290560 | 2.378813977
  EC-GC-2, CFAP54 | 1.988387042
  EC-GC-2, ABI3BP | 1.57362138
  EC-GC-2, SPACA6 | -1.724379529
  EC-GC-2, ADAMTSL2 | -2.009897896
  EC-GC-2, LZTS1 | -2.659531511
  EC-GC-2, ENSG00000285744 | 1.889210245
  EC-GC-2, ENSG00000225689 | -1.414674941
  EC-GC-2, LUZP2 | -4.384000321
  EC-GC-2, NCKAP5 | -1.592351284
  EC-GC-2, FAT1 | -1.855192898
  NKC-NKT, AGBL4 | -2.145446805
  NKC-NKT, TFEC | 1.989578132
  NKC-NKT, ENSG00000254186 | -2.913048038
  NKC-NKT, PDE10A | -2.170777761
  NKC-NKT, SHANK2 | -2.431773845
  PEC, RGS6 | -3.331377896
  PEC, AHNAK | -1.645129407
  PT-2, LRRC4C | -2.167101922
  PT-2, DSCAM | -3.104786855
  PT-2, RCN3 | -1.636040003

7. Secondary Outcome: Change in Glomerular Basement Membrane Width (Kidney Biopsy)
Description: Change in glomerular basement membrane width assessed in kidney biopsy from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Nanometer (nm)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 12 | 9
Nanometer (nm) | -72.67 (96.60) | -8.66 (206.35)

8. Secondary Outcome: Change in Apparent Diffusion Coefficient (ADC) (Cortex) (MRI)
Description: Change in apparent diffusion coefficient in cortex assessed by MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ADC (cortex)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of ADC (cortex)
  Bilateral cortex: number analyzed (Participants) | 51 | 29
  Bilateral cortex | 1.00 (6.56) | 0.94 (11.40)
  Left cortex: number analyzed (Participants) | 52 | 27
  Left cortex | 1.01 (8.50) | 0.96 (10.48)
  Right cortex: number analyzed (Participants) | 52 | 29
  Right cortex | 0.98 (6.70) | 0.93 (12.12)

9. Secondary Outcome: Change in Apparent Diffusion Coefficient (ADC) (Medulla) (MRI)
Description: Change in apparent diffusion coefficient in medulla assessed by MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ADC (medulla)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of ADC (medulla)
  Bilateral medulla: number analyzed (Participants) | 50 | 29
  Bilateral medulla | 0.98 (8.90) | 0.94 (13.51)
  Left medulla: number analyzed (Participants) | 52 | 27
  Left medulla | 0.99 (9.51) | 0.95 (13.41)
  Right medulla: number analyzed (Participants) | 51 | 29
  Right medulla | 0.98 (10.00) | 0.93 (13.94)

10. Secondary Outcome: Change in Mean Renal Artery Resistive Index (RARI) (MRI)
Description: Change in renal arterial resistive index assessed by MRI from baseline (week 0) to end of treatment (week 52) is presented. RARI measures the preservation of blood flow in renal arteries throughout the cardiac cycle and is therefore a measure for resistance of blood flow within the renal arteries. It serves as an indicator of kidney vascular health and potential arterial stiffness or obstruction. It is prognostic for primary cardiovascular and renal events in type 2 diabetes, where a lower RARI predicts a lower rate of events. RARI is calculated by relating the difference between blood flow at maximum velocity during the cardiac contraction phase (peak systolic velocity, PSV) and the speed at the end of the relaxation phase, at the point of minimal velocity (end diastolic velocity, EDV) with PSV, i.e., RARI = (PSV-EDV)/PSV.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of RARI
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of RARI
  Bilateral renalartery: number analyzed (Participants) | 54 | 32
  Bilateral renalartery | 0.97 (7.00) | 1.01 (6.13)
  Right renalartery: number analyzed (Participants) | 56 | 33
  Right renalartery | 0.98 (8.38) | 1.01 (8.62)
  Left renalartery: number analyzed (Participants) | 55 | 30
  Left renalartery | 0.97 (7.44) | 1.01 (6.43)

11. Secondary Outcome: Change in Mean Arterial Flow (MRI)
Description: Change in mean arterial flow assessed by MRI from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of mean arterial flow
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 71 | 35
Ratio of mean arterial flow
  Bilateral renalartery: number analyzed (Participants) | 56 | 32
  Bilateral renalartery | 0.96 (24.96) | 0.96 (25.06)
  Right renalartery: number analyzed (Participants) | 56 | 33
  Right renalartery | 0.97 (30.21) | 0.95 (29.09)
  Left renalartery: number analyzed (Participants) | 57 | 30
  Left renalartery | 0.96 (25.06) | 0.98 (27.38)

12. Secondary Outcome: Change in Natriuresis (Urinary Sodium Excretion) (Urinalysis)
Description: Change in natriuresis (urinary sodium excretion) (urinalysis) from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per day (mmol/day)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 57 | 32
Millimoles per day (mmol/day) | -7.3 (71.3) | -26.9 (85.2)

13. Secondary Outcome: Change in Albumin Excretion Rate (Urinalysis)
Description: Change in albumin excretion rate (urinalysis) from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milligrams per day (mg/d)
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 56 | 33
Milligrams per day (mg/d) | -81.9 (708.8) | -233.2 (964.8)

14. Secondary Outcome: Change in Kidney Function (Creatinine Clearance) (Urinalysis)
Description: Change in kidney function (creatinine clearance) (urinalysis) from baseline (week 0) to end of treatment (week 52) is presented.
Time Frame: Baseline (week 0), End of treatment (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 53 | 33
Milliliter per minute | 3.8 (26.6) | -12.6 (34.2)

ADVERSE EVENTS:
Time Frame: Up to week 57
Description: Safety analysis set- all participants randomly assigned to trial treatment & who take at least 1 dose of trial product. All presented AEs are treatment emergent adverse events (TEAEs). A TEAE was defined as an AE with onset in all observed data points from first date of study product until permanent discontinuation of treatment. A participant died after discontinuing study by physician decision hence was counted in 'physician decision' category in 'Participant Flow' in semaglutide arm.
Arm/Group | Semaglutide 1.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/71 | 1/35
Serious Adverse Events (participants affected / at risk) | 14/71 | 5/35
Other Adverse Events (participants affected / at risk) | 15/71 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=71) | Placebo (N=35)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=71) | Placebo (N=35)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04865770/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04865770/SAP_001.pdf